CLINICAL TRIAL: NCT03976765
Title: Early Rehabilitation Program in Liver Transplant Surgery: Hospital Discharge at Day 7 in a Targeted Population
Brief Title: Interest of an Early Rehabilitation Program in Liver Transplant Surgery
Acronym: RAC-TH
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_9723_RAC-TH
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital discharge at day 7
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — The patients follow different rehabilitation programs (surgery, anesthetic, post-operative). Hospital discharge is authorized only after validation of objective, clinical and para clinic criteria

SUMMARY:
Monocentric, prospective study to evaluate 10 liver transplanted patients

DETAILED DESCRIPTION:
The improvement of perioperative technics and the prevention of complications with immunosuppression allowed for the development with success of liver transplant. 1322 liver transplants occurred in 2016 in France to 806 in 2000. Centre Hospitalier Universitaire (CHU) of Rennes became a reference with 122 liver transplants in 2016 being the second liver transplant center in France.

Early rehabilitation concept is a multidisciplinary approach (surgical, anesthetic…) that aims to reduce the length of hospital stay and peri operative morbidity/mortality. These programs have first been developed in colorectal surgery before extending to complicated surgery like cephalic duodeno-pancreatectomy or hepatectomy. There are poor data in the literature on early rehabilitation program in liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* First liver transplant
* Liver transplant alone
* MELD (Model for End stage Liver Disease) score ≤ 15
* CHILD-PUGH score ≤ 8 if cirrhosis
* Body Mass Index < 30 kg/m2
* No history of transplant nor immunosuppression
* Absence of ascites nor hydrothorax drain
* Absence of treatment for diabetes
* Absence of renal insufficiency (glomerular filtration flow > 60 mL/min)
* Family help at home

Exclusion Criteria:

* Cold ischemia time > 8 hours
* Grafts from type III Maastricht
* Super urgent liver transplantation
* Perioperative blood transfusion > 4 packed red blood cells and/or 3 fresh frozen plasma
* Arterial anastomosis in splenic artery, in aorta or in coeliac artery
* Bilio-digestive anastomosis
* Persons deprived of liberty
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with an hospital discharge at day 7 | Day 7

SECONDARY OUTCOMES:
Number of patients readmission in the first month | Month 1
Number of days of hospitalization during the first month (post-surgery and prehospitalization) | Month 1
Number of death in the first month | Month 1
Satisfaction of the patient in the first month | Month 1
Number of surgery complications according to Dindo and Clavien classification during the first month | Month 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No